CLINICAL TRIAL: NCT02765282
Title: Automated Deep Brain Stimulation Programming Using Functional Mapping
Acronym: DBS-Expert
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: Wake Forest University Health Sciences (Other); Ohio State University (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: R44NS081902 (NIH)
Record Dates: First submitted 2016-04-27; First posted 2016-05-06 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation (DBS); Kinesia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DBS-Expert Programming First (Experimental): These patients will be undergo algorithm based programming using Kinesia-based assessment (DBS-Expert) first and then be programmed by a clinician within five days.
  Interventions: Device: Algorithm based programming using Kinesia-based assessment
- Traditional Programming First (Experimental): These patients will be programmed by a clinician first and then undergo algorithm based programming using Kinesia-based assessment (DBS-Expert) within five days.
  Interventions: Device: Algorithm based programming using Kinesia-based assessment

INTERVENTIONS:
Device: Algorithm based programming using Kinesia-based assessment — DBS-Expert includes a tablet-based software application (app) for guiding DBS programming and a Kinesia motion sensor unit for automated motor assessment. Algorithms search the programming parameter space to resolve an optimal set of programming parameters.
  Other Names: DBS-Expert

SUMMARY:
Participants will undergo DBS programming guided by the DBS-Expert system and by a clinician per standard care.

ELIGIBILITY:
Inclusion Criteria:

* The ability to provide informed consent
* Clinical diagnosis of idiopathic Parkinson's disease (PD)
* Implanted deep brain stimulation (DBS) system for tremor and/or bradykinesia

Exclusion Criteria:

* Significant medical or psychiatric illness or dementia as evidenced by a score less than 26 on the Montreal Cognitive Assessment
* Not capable of functioning independently
* Individuals so symptomatic as to compromise safety

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Programming time when programmed using Kinesia-based assessment (DBS-Expert) compared to programming time when programmed by a clinician | Up to 2 hours (from start of programming session until end of programming session)
  Amount of time it took to arrive at DBS settings that provide sufficient therapeutic benefit will be compared across programming sessions

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (3):
- United States (3):
  - Atrium Health, Charlotte, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio